CLINICAL TRIAL: NCT02680236
Title: Can Art Therapy Improve Breast Cancer Patients' Perception of Persistent Post Treatment Pain and Functioning? A Mixed Methods Pilot Study
Brief Title: Art Therapy for Pain Relief in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4218
Record Dates: First submitted 2016-01-05; First posted 2016-02-11 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: Pain; Cancer; Chemotherapy; Anxiety; Depression; Isolation
MeSH Terms: conditions — Pain; Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: This pilot study proposes to explore the effect of art therapy on breast cancer patients' perception of pain, and its impact on daily functioning by offering four sessions of individual art therapy, spaced between one to three weeks apart.
  The study will be open to breast cancer patients over the age of 18, who have been assessed by the Royal Marsden (RM) Pain Team, and who report having persistent post treatment pain of at least moderate intensity for the preceding two weeks despite having been optimally treated for their pain already, and who fulfil the inclusion criteria.
  Interventions: Other: Art Therapy Group

INTERVENTIONS:
Other: Art Therapy Group — Patients fulfilling the inclusion criteria will be made an appointment with the art therapist for the Initial Assessment session. They will be given the following Reflect Interview session Final interview session An analgesic use form will be given to the patient to take home to note their actual analgesic use
  At the end of each of these art therapy sessions, patients will be given a Brief Pain Inventory form (BPI) with a stamped addressed envelope. This is to be completed twenty four hours after the appointment and returned by post.

SUMMARY:
Art therapy offers benefits and support for a range of psychological symptoms caused by cancer and its treatments, for example anxiety, stress, depression, sleeplessness, identity or end of life concerns. Persistent post treatment pain that adversely affects quality of life may be experienced by up to 50% of breast cancer patients. Factors such as depression, fear, anxiety or lack of sleep are shown to increase pain and suffering in people with cancer. A multitreatment approach treatment of cancer pain is therefore recommended. Art therapy offers an opportunity to communicate the experience of suffering in a non verbal mode and can be offered in addition to other treatment for pain. This pilot study proposes to explore the effect of art therapy on breast cancer patients' perception of pain, and its impact on daily functioning by offering four sessions of individual art therapy, spaced between one to three weeks apart.

DETAILED DESCRIPTION:
Art therapy is a type of psychotherapy that uses making art and creative processes to allow patients to express feelings that may be difficult to put into words. It has been available at The Royal Marsden NHS Foundation Trust since 1988. Patients are referred for a range of issues that include isolation, anxiety, depression, identity or end of life issues. Research has shown art therapy to offer significant improvements in these areas. There is much anecdotal evidence within art therapy of it's effectiveness for physical pain, but little research in this area. Pain itself is acknowledged as a complex phenomena that demands a multifocused approach to treatment. The British Pain Society's guidelines recommend a combined approach to treatment that includes psychological and complementary therapies, but although music therapy is cited, art therapy is not. This study proposes to broaden the research base into art therapy's effectiveness as an additional intervention to support patients managing physical pain, and thus be able to be offered as additional support to the interventions currently on offer.

Art therapy would, in practice be able to be offered concurrently to all other treatments for pain, and at at any point in the treatment journey. However for the purpose of this study, in order to understand art therapy's potential effectiveness, it is useful to narrow the focus of the research. It is reported that up to 50% of breast cancer patients suffer from chronic post treatment pain, that is, for an extended period of time after all treatment for cancer and despite being optimally treated already for their pain. In consultation with the Pain Team at the RM it was decided that breast cancer patients were a suitable cohort for this study.

As this is the first study at the RM looking into art therapy and physical pain, it was decided that a mixed method study would produce the most valuable data. Narrative data from interviews will allow a greater understanding of participants experience of art therapy, and how it might be effective for pain. Numerical data will give information on the extent of how effective for pain art therapy might be. The sample size is small (20 participants) in order to allow for in depth analysis of the narrative data. Previous research studies looking at art therapy in oncology have offered between a single, to eight, one hour individual art therapy sessions. Art therapy research in oncology that included pain as a criteria for study, has offered a single, hour long session and examined data on its impact on pain collected immediately after the art therapy session. As this study proposes to explore art therapy as an intervention that may offer benefits for pain that develop over time, four, hour long individual art therapy sessions have been decided on. This allows for an understanding of whether art therapy may have any effect on pain beyond an immediate lessening during an art therapy session.

ELIGIBILITY:
Inclusion Criteria:

* reporting pain of longer than three months duration post chemotherapy, surgical or radiation treatment
* aged 18 years or older
* with more than two months predicted life expectancy
* who has English fluency
* who has capacity to consent
* wishing to access art therapy
* who is assessed by the pain team as stable on their current medication

Exclusion Criteria:

* who is less than three months post their chemotherapy or radiation treatment, or who receives new chemotherapy or radiation treatment during the study.
* who has had pain reduction surgery less than three months before the study, or receives it during the study period
* who has had any change in medication for pain control less than two weeks prior to the study, or during the study period
* who scores less than moderate pain (less than 4 on a scale of 1 -10) in a verbal self-reported measure of their worst pain felt, for the preceding two weeks before the study period
* who intends to access art therapy outside the sessions offered within the study, for the duration of the study
* who receives other psychological therapies from another practitioner during the study period
* who receives physiotherapy for problems related to their breast cancer treatment during the study period
* who receives massage or reflexology treatments from the complementary therapy team during the study period

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with breast cancer as assessed by the RM pain team.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patient showing change in Brief Pain Inventory pain interference score | From baseline to end of the study (approx six months)
  The percentage of patients who will demonstrate a 2 point change in Brief Pain Inventory pain interference score from baseline to end of study.

SECONDARY OUTCOMES:
Percentage of patient showing change in Brief Pain Inventory pain severity score | From baseline to end of the study (approx six months)
  The percentage of patients who will demonstrate a 2 point change in Brief Pain Inventory pain severity score from baseline to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, BSc,RD,PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No